CLINICAL TRIAL: NCT06825130
Title: Feasibility and Preliminary Efficacy of High-intensity Interval Training Combined with Muscle-strength Training in Older Women: Pilot Randomized Controlled Trial
Brief Title: High-intensity Interval Training Combined with Muscle-strength Training in Older Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Tasuku Terada, Dr, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMHS 34-1124
Record Dates: First submitted 2025-02-03; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Older Adult
Keywords: Women; HIIT; Resistance exercise; Combined exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aerobic training + muscle strength training (Experimental): 3 days/week -- 3-min warm up at 60% of HR@VT2 on a bike ergometer -- 6 x 1-min machine-base muscle strength exercises: leg press, chest press, knee extension, lat pull down, knee flexion, and shoulder raise -- 6 x 1-min high-intensity interval bouts at 80% HR@VT2 interspersed by 1-min active recovery will be performed.
  Interventions: Behavioral: Exercise
- aerobic training (Active Comparator): 3 days/week -- 3-min warm up at 60% of HR@VT2 on a bike ergometer -- 2 blocks of 6 x 1-min high-intensity interval bouts at 70% HR@VT2 interspersed by 1-min active recovery
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will attend 30-min training sessions 3 times a week for 12 weeks. The intensity of HIIT will be at 80% HR@VT2 measured in the first week and will increase to 90% in the second week. By week 3, the intensity will reach HR@VT2.

SUMMARY:
Women generally live longer than men but often experience a faster muscle mass loss due to inactivity, which can lead to weakness and disability. Despite these risks, women, particularly older women, are less active than men. In England, less than one-third of women engage in sufficient aerobic activity, and less than 5% do enough muscle strength training. Common reasons for not exercising include lack of time and enjoyment.

High-intensity interval training (HIIT) is an efficient and effective way to exercise that many women find more enjoyable than longer workouts. HIIT has been shown to be effective in older women, helping them improve their fitness with less time commitment. Because HIIT is time-efficient, it can be combined with muscle strength training without significantly increasing the duration of the exercise session, which may lead to even better fitness results.

This study will assess how practical it is for older women to do HIIT and strength exercise combined training. It will also investigate whether this combined approach can improve overall fitness, muscle strength, aerobic fitness, and quality of life more than HIIT alone.

ELIGIBILITY:
Inclusion Criteria:

* Females (biologically at birth)
* At least 60 years of age at the time of signing the informed consent
* Non-smoker, including electronic cigarettes
* Not participating in routine high-intensity aerobic or muscle strength exercise training (≥ 75 min/week of structured vigorous aerobic exercise, or 2 times /week of structured muscle strength training)
* Able to perform a cardiopulmonary exercise testing (CPET) to exhaustion
* willing to complete baseline and follow-up measures, and attend prescribed exercise sessions at the University of Nottingham
* willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Diagnosed with cardiovascular disease, kidney disease, diabetes, obstructive pulmonary disease, or uncontrolled hypertension
* History or current neurological or psychiatric illness, or motor or cognitive restrictions
* Contraindications to symptom-limited cardiopulmonary exercise testing (CPET), including resting hypertension with systolic blood pressure >200 mmHg or diastolic blood pressure > 110 mmHg, uncorrected medical conditions, such as significant anemia, important electrolyte imbalance, and hyperthyroidism, mental impairment with limited ability to cooperate, physical disability that precludes safe and adequate testing.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of high-intensity interval training combined with muscle strength training | From recruitment to week-12
  will be assessed from recruitment, adherence, compliance, safety, subjective exercise experiences and self-efficacy. Recruitment will be assessed by the proportion of patients remained interested and randomized after being informed of the requirements of the study; adherence will be assessed by the attendance to the prescribed exercise sessions; and compliance will be assessed by the proportion of participants adhering to prescribed exercise intensity. For safety, all mild, moderate, and severe symptoms and adverse events throughout this study will be recorded.

SECONDARY OUTCOMES:
functional capacity | From baseline to week-12
  will be assessed using the Fullerton Functional Fitness Test, a valid and reliable measure of functional independence in older adults
muscle function | From baseline to week-12
  Isometric strength, isokinetic muscle torque (i.e., strength) and fatigue will be measured using a dynamometer (CYBEX).
cardiorespiratory fitness | From baseline to week-12
  will be measured by a gold-standard, symptom-limited CPET using metabolic equipment on an electronically braked cycle ergometer.
muscle mass | From baseline to week-12
  will be measured using ultrasound at the mind-point of the thigh, from the greater trochanter to mid patella.
QoL | From baseline to week-12
  will be assessed using Short Form 36 Health Survey Questionnaire (SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- David Greenfield Humnn Physiology Unit (DGHPU), University of Nottingham, Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided